CLINICAL TRIAL: NCT06534866
Title: "Effects of Kinesio Taping in Adjunct to Traditional Physical Therapy on Pain, Range of Motion and Gait Parameters in Patients With Plantar Fascitis : a Randomized Controlled Trail"
Brief Title: "Effects of Kinesio Taping in Adjunct to Traditional Physical Therapy on Pain, Range of Motion and Gait Parameters in Patients With Plantar Fasciitis : a Randomized Controlled Trail"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/23
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physcial therapy group (Active Comparator): 1. TENS+cold pack (For 10 mins on plantar ascpect of foot)
  2. Stretching exercises (5 repetition 2 sets/day) Standing calf stretch Seated plantar fascia stretch Plantar fascia massage Achilles stretch Frozen can roll Towel stretch (30 minutes session thrice a week for 2 consecutive weeks with total of 6 sessions)
  Interventions: Other: Traditional Physical Therapy
- Kinesio taping + Traditional physical therapy group (Experimental): Group B will receive :
  1. TENS+cold pack For 10 mins on plantar ascpect of foot
  2. Stretching exercises (5 repetition 2 sets/day) Standing calf stretch Seated plantar fascia stretch Plantar fascia massage Achilles stretch Frozen can roll Towel stretch
  3. Kinesio taping:
  (30 minutes session thrice a week for 2 consecutive weeks with total of 6 sessions)
  Interventions: Other: Traditional Physical Therapy; Other: Kinesiotaping

INTERVENTIONS:
Other: Traditional Physical Therapy — 1. TENS+cold pack (For 10 mins on plantar ascpect of foot)
  2. Stretching exercises (5 repetition 2 sets/day) Standing calf stretch Seated plantar fascia stretch Plantar fascia massage Achilles stretch Frozen can roll Towel stretch
Other: Kinesiotaping — In the first step, after the metatarsophalangeal joints is dorsiflexed, the first strap will be adhered firmly to the posterior heel at its proximal end. The other end of the strap is cut into four slices of equal width. Each slice is applied with a 50% stretch (50% tensile strain) and attached to the plantar forefoot. In the second step, another strap is applied with gentle compression across the bases of the four slices beneath the foot and wrapped around the rearfoot
  Arms: Kinesio taping + Traditional physical therapy group

SUMMARY:
THIS STUDY IS A RANDOMIZED CONTROL TRIAL AND THE PURPOSE OF THIS STUDY IS TO DETERMINE THE EFFECTS OF KINESIO TAPING ON GAIT PARAMETERS IN PATIENTS WITH PLANTAR FASCITIS

DETAILED DESCRIPTION:
The purpose of this study is to determine the difference between efffects of KInesio taping combined with traditional physical versus physical therapy alone.

The individual of Age 20-40 years among both genders and are diagnosed cases of plantar fasciitis Pain levels will be assessed using the Numeric Pain Rating Scale (NPRS). ROM will be assessed through goniometry. Gait parameters will be assessed through 30 meter walk test. Participants of interest would be approached and explained about the research. Informed written consent will be taken. It is a single-blinded study and randomization will be done through coin toss method. Both groups will receive conventional intervention. Additionally, Group B will receive kinesio taping treatment. Baseline and post intervention scores would be recorded for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 20-40 years
* Diagnosed Cases of plantar fasciitis as per diagnosis criteria established by APTA

As described by American Physical Therapy Association:

Plantar medial heel pain: most noticeable with initial steps after a period of inactivity but also worse following prolonged weight bearing

* Heel pain precipitated by a recent increase in weight-bearing activity
* Pain with palpation of the proximal insertion of the plantar fascia
* Positive windlass test
* Negative tarsal tunnel tests
* Limited active and passive talocrural joint dorsiflexion range of motion
* Abnormal Foot Posture Index score

Exclusion criteria:

* Recent steroid injections
* History of ankle or foot surgery
* Arthritis history
* Radiculopathy
* Diabetic foot

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 2 weeks
  Pain is assessed by using numeric main rating scale comparing pre and post pain intensity. This is 11- point numeric scale ranges from '0' representing one pain extreme (e.g., "no pain") to '10' representing the other pain extreme
Range of Motion at ankle joint | 2 weeks
  Goniometer will be used to measure the pre and post treatment ranges of dorsiflexion and plantar flexion of ankle in supine and sitting positions.
Cadence (steps/min) | 2 weeks
  Will asses gait parameters through 30 meters walk test. steps counted x 60 / time (s)
Cycle time (s) | 2 weeks
  Will asses gait parameters through 30 meters walk test. time (s) x 2/steps counted
Gait speed | 2 weeks
  Will asses gait parameters through 30 meters walk test. Distance (m) /time (s)
Stride length(m) | 2 weeks
  Will asses gait parameters through 30 meters walk test. speed (m/s) x cycle time (s)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan